CLINICAL TRIAL: NCT06515028
Title: The Effects of General Anesthesia and Infraclavicular Block Applications on Oxidative Stress and Endothelial Dysfunction in Upper Extremity Surgeries
Brief Title: Effects of Anesthesia Technique on Endothelial Function
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Sezen Kumaş Solak, Principle Investigator, Bagcilar Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Bagcılar2
Record Dates: First submitted 2024-07-10; First posted 2024-07-23 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Endothelial Dysfunction; Ischemia Reperfusion; Oxidative Stress
Keywords: endothelial dysfunction; ischemia reperfusion; oxidative stress; infraclavicular block; general anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group GA: general anesthesia (Active Comparator): Group GA
  Interventions: Procedure: Group GA
- Group IB : infraclavicular block (Active Comparator): Group IB
  Interventions: Procedure: Group IB

INTERVENTIONS:
Procedure: Group GA — Anesthesia induction will be performed preoxygenation with 3 minutes of 80% FiO2 , followed by intravenosus propofol 2-2.5 mg/kg and fentanyl 2 µg/kg. Rocuronium 0.6 mg/kg will be administered for neuromuscular blockade, followed by endotracheal intubation after 2 minutes of mask ventilation. Anesthesia maintenance will be achieved with inhalation of 2.5-3.3% sevoflurane with 50% oxygen and 50% air mixture, along with infusion of remifentanil at 0.1 micrograms/kg/min. ventilation will be performed using a volume-controlled.
  Arms: Group GA: general anesthesia
Procedure: Group IB — infraclavicular brachial plexus block will be performed in supine position with the arm adducted and flexed at 90 degrees. A mixture consisting of 15 ml of 0.5% Bupivacaine, 15 ml of 2% Lidocaine, and 30 ml of saline solution will be prepared, with equal concentrations distributed into three different syringes of 20 milliliters each. The clavicular notch will be palpated, and an ultrasound linear probe covered with a sterile sheath will be positioned in the lateral sagittal plane over this area to visualize the median, lateral, and posterior cords of the brachial plexus surrounding the axillary artery. A special Stimuplex A 22G, 100 mm needle will be used for plexus anesthesia. local anesthetic injection will be sequentially performed around the posterior, median, and lateral cords under ultrasound guidance. After confirming sensory and motor block, the operation will be commenced.
  Arms: Group IB : infraclavicular block

SUMMARY:
The aim of this study was to compare the effects of two different anesthesia methods, general anesthesia and infraclavicular block, on oxidative stress and endothelial dysfunction in upper extremity forearm operations.This prospective study aims to determine the ideal anesthesia method for patients undergoing upper extremity forearm surgeries under tourniquet by comparing general anesthesia and infraclavicular block applications in terms of oxidative stress and ED related to ischemia-reperfusion injury.

DETAILED DESCRIPTION:
Pneumatic tourniquets are commonly used in orthopedic extremity surgeries to reduce surgical trauma and blood loss. When the tourniquet is released, it leads to the release of more free oxygen radicals than under physiological conditions, resulting in ischemia-reperfusion injury, oxidative stress, and endothelial dysfunction (ED).

Endothelial dysfunction is characterized by the imbalance between vasoactive substances such as nitric oxide (NO) and endothelin, which regulate vascular tone by exerting vasodilatory and vasoconstrictive effects.During ischemia, xanthine oxidase (XO) derived from xanthine dehydrogenase is the main source of free oxygen radicals (FOR), including superoxide anion (O2-), hydrogen peroxide (H2O2), and hydroxyl anion (OH-). Superoxide anion reacts with NO to produce peroxynitrite (ONOO-), a reactive oxygen derivative. Free radicals affect unsaturated fatty acids in membranes, leading to the production of malondialdehyde (MDA), which exerts cytotoxic effects on endothelial cells. Increased production of FOR due to oxidative stress and dysfunction of antioxidant mechanisms result in protein carbonylation. Protein carbonyl groups (PC) serve as indicators of severe oxidative damage and loss of protein function

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for upper extremity surgery using a pneumatic tourniquet
* American Society of Anesthesiologists (ASA) physical status classification I

Exclusion Criteria:

* Under 18 or over 65 years of age
* Hypertension
* Diabetes mellitus
* Malignancy
* Cardiovascular disease history (congestive heart failure, myocardial infarction, venous thrombosis)
* Cerebrovascular disease history
* Liver/kidney dysfunction
* Pregnant or breastfeeding women
* History of substance and tobacco use
* History of extremity ischemia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2024-08-25 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Effects of Anesthesia Technique on Endothelial Function with using ultrasonographic technique | Brachial artery FMD measurements will evaluated using ultrasonographic technique from the contralateral Measurements will be taken at three different time points: preoperatively(FMD1), 24hours postoperatively (FMD2), 6th day postoperatively(FMD3)
  In this study, investigators aimed to determine the ideal anesthesia method for patients undergoing upper extremity surgeries accompanied by a tourniquet, by comparing general anesthesia and infraclavicular block methods in terms of oxidative stress and endothelial dysfunction (ED) related to ischemia-reperfusion injury. Brachial artery FMD (flow-mediated dilation ) measurements will evaluated using ultrasonographic technique from the contralateral
Evaluation of the Effect of Anesthesia Technique on Endothelial Function with evaluated in the collected blood samples levels | before anesthesia (T0), 1 minute before (T1), 5 minutes after (T2), and 20 minutes after deflation of the tourniquet
  During the operation, the dorsal venous cannula in the foot was not utilized for any other purpose. The duration of surgery and tourniquet application was recorded for each group. Tourniquet pressure was set at approximately twice the systolic arterial pressure (SAP). Evaluated in the collected blood samples levels of Protein carbonyl (PC),xanthine oxidase (XO),nitric oxide (NO),malondialdehyde (MDA)

SECONDARY OUTCOMES:
Effects of Anesthesia Technique on Endothelial Function | before anesthesia (T0), 1 minute before (T1), 5 minutes after (T2), and 20 minutes after deflation of the tourniquet
  During the operation, the dorsal venous cannula in the foot was not utilized for any other purpose. The duration of surgery and tourniquet application was recorded for each group. Tourniquet pressure was set at approximately twice the systolic arterial pressure (SAP). SAP, diastolic arterial pressure (DAP), mean arterial pressure (MAP), and heart rate (HR) values were recorded at time points T0, T1, T2, and T3.

CONTACTS AND LOCATIONS:
Overall Officials: SEZEN KUMAS SOLAK, Principal Investigator — Bagcılar Training Research Hospital

IPD SHARING:
Plan to Share IPD: No
The investigators will not share individual patient data

REFERENCES:
- [Background] Rosenfeldt F, Wilson M, Lee G, Kure C, Ou R, Braun L, de Haan J. Oxidative stress in surgery in an ageing population: pathophysiology and therapy. Exp Gerontol. 2013 Jan;48(1):45-54. doi: 10.1016/j.exger.2012.03.010. Epub 2012 Mar 23. PMID 22465624
- [Background] Gourdin MJ, Bree B, De Kock M. The impact of ischaemia-reperfusion on the blood vessel. Eur J Anaesthesiol. 2009 Jul;26(7):537-47. doi: 10.1097/EJA.0b013e328324b7c2. PMID 19412112
- [Background] Vlachopoulos C, Xaplanteris P, Aboyans V, Brodmann M, Cifkova R, Cosentino F, De Carlo M, Gallino A, Landmesser U, Laurent S, Lekakis J, Mikhailidis DP, Naka KK, Protogerou AD, Rizzoni D, Schmidt-Trucksass A, Van Bortel L, Weber T, Yamashina A, Zimlichman R, Boutouyrie P, Cockcroft J, O'Rourke M, Park JB, Schillaci G, Sillesen H, Townsend RR. The role of vascular biomarkers for primary and secondary prevention. A position paper from the European Society of Cardiology Working Group on peripheral circulation: Endorsed by the Association for Research into Arterial Structure and Physiology (ARTERY) Society. Atherosclerosis. 2015 Aug;241(2):507-32. doi: 10.1016/j.atherosclerosis.2015.05.007. Epub 2015 May 16. PMID 26117398